CLINICAL TRIAL: NCT01464554
Title: Brief Substance Use Intervention for Youth in Teen Court
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA019938-01 (NIH)
Record Dates: First submitted 2011-07-20; First posted 2011-11-03 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Alcohol or Other Drugs Use
Keywords: adolescents; alcohol; drugs; delinquency; intervention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Teens will receive six sessions of an alcohol and drug education group
  Interventions: Behavioral: Usual care
- Project Free Talk (Experimental): Teens will receive six sessions of and evidenced based motivational interviewing alcohol and drug program
  Interventions: Behavioral: Project Free Talk

INTERVENTIONS:
Behavioral: Usual care — alcohol and drug education
  Other Names: ADAG
  Arms: Usual Care
Behavioral: Project Free Talk — motivational interviewing alcohol and drug program
  Arms: Project Free Talk

SUMMARY:
Youth involved in the juvenile justice system have multiple problems, including an earlier onset of alcohol and drug use and higher rates of alcohol and drug use than their peers in the general population. This 4.5 year study will develop and evaluate a new group intervention for youth who have committed a first time alcohol or drug offense. Teens will be randomized to receive either usual care or the new group intervention. Teens will complete a baseline, post-test (when they complete the intervention, which could vary for each teen but is typically around 6-8 weeks), and a 3-month follow-up survey upon completion of the intervention. The investigators will examine outcomes for a variety of behaviors, including alcohol and drug use and assess whether there are differences between the teens who received usual care and the teens who received the new group intervention.

DETAILED DESCRIPTION:
It is well known that youth involved in the juvenile justice system have multiple problems, including an earlier onset of alcohol and drug use and higher rates of alcohol and drug use than their peers in the general population. Several recent innovative treatment approaches have been developed to address substance use and the multiple problems that these at-risk youth experience. What is less well documented, however, are innovative approaches to treat youth who are first time alcohol or drug offenders and who may just be beginning to experience problems due to their substance use. The investigators propose a 4.5 year study to adapt and test an efficacious group intervention among teens who have committed a first time alcohol or other drug misdemeanor offense. These teens have been referred by the juvenile Probation Department to a Teen Court program because they have not been found to need more serious intervention such as treatment or detention. The objectives of the proposed research are to: Aim 1. Design a developmentally sensitive intervention curriculum in which the investigators (a) utilize our previous work and components from relevant existing approaches targeting at-risk adolescents, (b) establish participant acceptance, and (c) establish feasibility of intervention delivery with the participants, providers and the proposed setting; Aim 2. Implement a pilot test of the revised intervention with an adolescent population of first time offenders in which the investigators (a) demonstrate our ability to retain sufficient numbers of this population; (b) ensure intervention fidelity throughout the course of the study and (c) evaluate participant satisfaction, group engagement, and group climate; Aim 3. Examine the impact of the intervention on cognitive and behavioral outcomes to determine (a) whether clinically significant changes in expectancies, perceived prevalence of peer use, self-change efforts, alcohol consumption, marijuana and other drug use, and related consequences occur; (b) if reductions occur, estimate the likely effect sizes, and (c) explore the mechanism of change for decreases in substance use and consequences through mediation analyses. Our study seeks to narrow the gap between research and practice and builds upon recommendations by NIDA's Blue Ribbon Task Force by conducting research in a nonacademic setting with a population at high risk for alcohol and drug abuse. This study will extend selective intervention research for at-risk youth, as it will be one of the first to examine the impact of a theoretically based selective intervention for first time juvenile Alcohol or Other Drug (AOD) offenders.

ELIGIBILITY:
Inclusion Criteria:

* 14-18 years old;
* English speaking

Exclusion Criteria:

* has medical marijuana card;
* is older or younger than 14-18 years old,
* does not speak English

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 193 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
frequency of alcohol and drug use | three month follow up
  this will include the frequency of drinking and the frequency of marijuana use

SECONDARY OUTCOMES:
frequency of other risk behaviors | 3 month follow up
  this will include sexual behavior and delinquent behavior

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. D'Amico, Ph.D., Principal Investigator — RAND
Locations (1):
- The Council on Drug and Alcohol Abuse, Santa Barbara, California, United States